CLINICAL TRIAL: NCT07299006
Title: Evaluation of Paro, a Therapeutic Assistance Robot in Analgesic Management During the Placement of a Peripheral Intravenous Line in Infants and Children, a Multicenter Randomized Prospective Study.
Brief Title: Evaluation of Paro, a Therapeutic Assistance Robot in Analgesic Management During the Placement of a Peripheral Intravenous Line in Infants and Children.
Acronym: PARO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 24-HPNCL-05 PARO; 2025-A00617-42 (Other: ANSM)
Record Dates: First submitted 2025-11-27; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group : standard multimodal stratgey (Active Comparator): The child will go to the emergency room. If EMLA cream is used to stop pain, it will be put on the skin 30 minutes to 1 hour before the procedure.
  If MEOPA is used to help with pain, the child will wear a mask with the gas. The procedure starts by cleaning the skin and finding a vein. The procedure really begins when the needle first goes into the skin. The procedure ends when the needle is taken out and a bandage is put on
  Interventions: Drug: non- pharmacological interventions and usual pharmacological interventions
- tes group: standard multimodal Strategy with PARO robot (Experimental): The child will be taken to the emergency room. If EMLA cream is used to reduce pain, it will be put on the skin 30 minutes to 1 hour before the procedure.
  To help the child feel comfortable with PARO, the robot will be placed on or next to the child's lap 15 minutes before the procedure starts.
  If MEOPA is used to relieve pain, the mask with the gas will be put on the child's face.
  The procedure will start with cleaning the skin and looking for a vein. The procedure officially begins when the skin is first pierced. The procedure will finish when the needle is taken out and a bandage is put on.
  Interventions: Device: Test group : standard multimodal strategy with PARO robot

INTERVENTIONS:
Device: Test group : standard multimodal strategy with PARO robot — The child will be taken to the emergency room. If EMLA cream is used to reduce pain, it will be put on the skin 30 minutes to 1 hour before the procedure.
  To help the child feel comfortable with PARO, the robot will be placed on or next to the child's lap 15 minutes before the procedure starts.
  If MEOPA is used to relieve pain, the mask with the gas will be put on the child's face.
  The procedure will start with cleaning the skin and looking for a vein. The procedure officially begins when the skin is first pierced. The procedure will finish when the needle is taken out and a bandage is put on.
  Arms: tes group: standard multimodal Strategy with PARO robot
Drug: non- pharmacological interventions and usual pharmacological interventions — Pharmacological therapies : EMONO and EMLA cream EMONO = Equimolar Mixture of Oxygen and Nitrous Oxide EMLA cream = Eutectic Mixture of Local Anesthetics cream Non-pharmacological interventions (include music therapy and watching cartoons).
  Arms: Control group : standard multimodal stratgey

SUMMARY:
Peripheral intravenous catheterization is one of the most frequently performed procedures in children in emergency rooms and pediatric units. It often causes anxiety for both the child and their parents, which increases the pain associated with the procedure itself, as fear and pain are closely linked. Managing the child's pain and anxiety is essential to optimize the child's well-being in the short, medium, and long term.

The quality of pediatric analgesia largely depends on the multimodal approach to interventions offered to children in pain. Recently, several non-pharmacological therapies for pain management and anxiety reduction have been developed. Among these techniques, new technologies have emerged, such as therapeutic assistance robots equipped with artificial intelligence, but their therapeutic benefits still need to be evaluated.

The investigators therefore aim to conduct a study on PARO, a therapeutic assistance robot shaped like a baby seal, to evaluate its role in pain management during peripheral venous catheterization in children. The investigators intend to compare the therapeutic effects of PARO combined with standard techniques versus standard techniques alone during painful procedures. The objective is to determine whether the use of this therapeutic assistance robot can improve and optimize the overall management of children undergoing needle-induced skin punctures. Thus, the investigators plan a multicenter, randomized, open-label, superiority study conducted in five pediatric centers. The investigators aim to recruit 120 infants and children aged 12 months to 7 years who will undergo peripheral venous catheterization. Pain will be assessed using the FLACC (Face-Legs-Activity-Cry-Consolability) hetero-assessment scale in this age group.

Secondary objectives include assessing and comparing distress in the two groups using the PRIC (Procedural Restraint Intensity for Children) tool, which measures restraint intensity, as well as monitoring heart rate variability, the number of attempts required to complete the procedure, parental anxiety via the STAI (State-Trait Anxiety Inventory) questionnaire, and finally, the satisfaction of both parents and paramedical staff.

ELIGIBILITY:
Inclusion Criteria:

1. are between 12 months and 7 years old
2. require a peripheral intravenous catheterization (PIC)
3. speak and understand French.

Exclusion Criteria:

1. the need for contact isolation including colonization or infection with multidrug-resistant bacteria (MRB),
2. visual or hearing impairment;
3. psychiatric pathology that could impair the understanding;
4. life-threatening emergency;
5. the requirement for stronger analgesic drugs (such as Morphine, Ketamine, and intranasal therapeutics).

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Pain assessed using the FLACC (Face-Legs-Activity-Cry-Consolability) scale. | periprocedural
  The effectiveness of PARO in reducing pain during the procedure will be assessed using the FLACC (Face-Legs-Activity-Cry-Consolability) hetero-evaluation scale. The FLACC is a validated hetero-assessment tool used for the evaluation of pain in children aged between 12 months and 7 years old, particulary in the immediate postoperative pain and during brief pain associated with medical procedures. This scale assesses five behavioral parameters: facial expression, leg movement, activity, crying, and consolability. Each parameter is scored from 0 to 2, resulting in a total score ranging from 0 to 10. A score of 0 indicates a relaxed and comfortable child, while scores between 7 and 10 reflect severe pain or significant distress. A score of 3 or above is considered to be the threshold for initiating pain treatment.

SECONDARY OUTCOMES:
Heart rate measure | periprocedural
  Heart rate variability serves as a physiological indicator of pain, reflecting changes in sympathetic and parasympathetic nervous system activity in response to nociceptive stimuli.
Parental anxiety assessment using the STAI (State Trait Anxiety Inventory) questionnaire. | at the end of the procedure
  Parental anxiety will be assessed using the STAI (State Trait Anxiety Inventory) questionnaire. The STAI is a self-administered questionnaire containing 40 items, divided into two subscales: one assessing state anxiety (AE), which reflects the current emotional state (STAI-form Y-1), making it possible to assess the patient's nervousness and anxiety; the other assessing trait anxiety (AT), which reflects the general or baseline level of anxiety (STAI-form Y-2). Each response to an item of the STAI is scored from 1 to 4, with 1 indicating the lowest degree of anxiety and 4 the highest degree.
failure rate of peripheral intravenous catheterization | periprocedural
  Failure is defined as the inability to establish a peripheral intravenous access after three attempts (as defined above), and the need to ask the anesthesia team to perform it.
questionnaire of Parental satisfaction | 15 minutes after the end of the procedure
  Parental satisfaction will be evaluated using a questionnaire given to parents. This questionnaire consists of four items with Lickert-type response scale.
Questionnaire of paramedical team satisfaction | 15 minutes after the end of the procedure.
  The satisfaction of the paramedical team will be assessed using a separate questionnaire. This questionnaire will be distributed to all nursing staff involved in the study upon its completion and will be completed only once by each participant. It consists of four items with Likert-type response scales. Additionally, one or more feedback meetings will be organized with the care team at the end of the study to discuss their experiences and opinions regarding the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara LE GALLO, MD, Principal Investigator — Hôpitaux pédiatrique Nice CHU Lenval
Locations (1):
- Fondation Lenval Hôpitaux pédiatrique Nice CHU Lenval, Nice, France

IPD SHARING:
Plan to Share IPD: No